CLINICAL TRIAL: NCT04338009
Title: The Randomized Elimination or Prolongation of Angiotensin Converting Enzyme Inhibitors and Angiotensin Receptor Blockers in Coronavirus Disease 2019
Brief Title: Elimination or Prolongation of ACE Inhibitors and ARB in Coronavirus Disease 2019
Acronym: REPLACECOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Jordana B. Cohen, MD, MSCE (Unknown); Hanff, Thomas C., M.D., MPH (Individual); University of Arizona (Other); Hospital Nacional Carlos Alberto Seguin Escobedo - EsSalud (Other); Hospital Nacional Edgardo Rebagliati Martins (Other); Hospital Español de Mendoza (Other); Stanford University (Other); Ottawa Hospital Research Institute (Other); Hospital Civil de Guadalajara (Other); Universidad Catolica Argentina (Other); Caja Nacional de Salud (Other); Departamento de Medicina, Hospital Alberto Barton Thompson, Callao, Peru (Other); Karolinska Institutet (Other); University of Miami (Other); Division of Cardiology, Department of Medicine, Hospital Español, Buenos Aires, Argentina (Other); University of Michigan (Other); Jesse Chittams, MS (Unknown); Duke University (Other); Vasquez, Charles R., M.D. (Individual)
Responsible Party: Principal Investigator, Julio A. Chirinos, Associate Professor of Medicine at the Hospital of the University of Pennsylvania, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 842810
Record Dates: First submitted 2020-04-01; First posted 2020-04-08 (Actual); Results first posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discontinuation arm (Experimental): The randomized intervention will be the discontinuation of ACEI/ARBs
  Interventions: Other: Discontinuation of ARB/ACEI
- Continuation arm (Experimental): The randomized intervention will be the continuation of ACEI/ARBs
  Interventions: Other: Continuation of ARB/ACEI

INTERVENTIONS:
Other: Discontinuation of ARB/ACEI — The randomized intervention will be the discontinuation of ACEI/ARBs. In all participants randomized to discontinuation, treating clinicians will be reminded about the medication discontinuation upon discharge and will be prompted to consider re-initiation of the medication at that time if appropriate, per the clinician's discretion.
  Arms: Discontinuation arm
Other: Continuation of ARB/ACEI — The randomized intervention will be the continuation of ACEI/ARBs at the doses previously prescribed for patients during their routine care. Clinicians will be encouraged to continue the randomized treatment but will be allowed to change the dose of ACEI/ARB or discontinue these medications if any compelling clinical reasons are identified (such as hypotension, hyperkalemia, acute kidney injury).
  Arms: Continuation arm

SUMMARY:
The severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the virus responsible for coronavirus disease 2019 (COVID-19), is associated with a high incidence of acute respiratory distress syndrome (ARDS) and death. Hypertension and cardiovascular disease are risk factors for death in COVID-19. Angiotensin converting enzyme 2 (ACE2), an important component of the renin-angiotensin system, serves as the binding site of SARS-CoV-2 and facilitates host cell entry in the lungs. In experimental models, angiotensin converting enzyme inhibitors (ACEIs) and angiotensin receptor blockers (ARBs) have been shown to increase ACE2 expression in several organs, potentially promoting viral cell invasion, although these findings are not consistent across studies. Alternatively, ACEIs and ARBs may actually improve mechanisms of host defense or hyperinflammation, ultimately reducing organ injury. Finally, ACEIs and ARBs may have direct renal, pulmonary and cardiac protective benefits in the setting of COVID-19. Therefore, it is unclear if ACEIs and ARBs may be beneficial or harmful in patients with COVID-19. Given the high prevalence of hypertension, cardiovascular and renal disease in the world, the high prevalence of ACEIs or ARBs in these conditions, and the clinical equipoise regarding the continuation vs. discontinuation of ACEIs/ARBs in the setting of COVID, a randomized trial is urgently needed. The aim of this trial is to assess the clinical impact of continuation vs. discontinuation of ACE inhibitors and angiotensin receptor blockers on outcomes in patients hospitalized with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Hospitalization with a suspected diagnosis of COVID-19, based on: (a) A compatible clinical presentation with a positive laboratory test for SARS-CoV-2, or (b) Considered by the primary team to be a Person Under Investigation due to undergo testing for COVID-19 in addition to compatible pulmonary infiltrates on chest x-ray (mutilobar, intersticial or ground glass opacities).
3. Use of ACEI or ARB as an outpatient prior to hospital admission.

Exclusion Criteria:

1. Systolic blood pressure <100 mmHg.
2. Systolic blood pressure > 180 mmHg or >160 if unable to substitute ACEIs/ARBs for another antihypertensive class, per the investigator's discretion.
3. Diastolic blood pressure > 110 mmHg
4. Known history of heart failure with reduced ejection fraction (EF <40%) on their most recent echo and/or clinical heart failure with unknown EF (i.e. no echo in approximately the past year).
5. Serum K>5.0 mEq/L on admission.
6. Known pregnancy or breastfeeding.
7. eGFR <30 mL/min/1.73m2
8. >50% increase in creatinine (to a creatinine >1.5 mg/dl) compared to most recent creatinine in the past six months, if available
9. Urine protein-to-creatitine ratio > 3 g/g or proteinuria > 3 g/24-hours within the past year
10. Ongoing treatment with aliskiren or sacubitril-valsartan.
11. Inability to obtain informed consent from patient.
12. Inability to read and write or lack of access to a smart phone, computer or tablet device at the time of evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Not making it available

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Forouzanfar MH, Liu P, Roth GA, Ng M, Biryukov S, Marczak L, Alexander L, Estep K, Hassen Abate K, Akinyemiju TF, Ali R, Alvis-Guzman N, Azzopardi P, Banerjee A, Barnighausen T, Basu A, Bekele T, Bennett DA, Biadgilign S, Catala-Lopez F, Feigin VL, Fernandes JC, Fischer F, Gebru AA, Gona P, Gupta R, Hankey GJ, Jonas JB, Judd SE, Khang YH, Khosravi A, Kim YJ, Kimokoti RW, Kokubo Y, Kolte D, Lopez A, Lotufo PA, Malekzadeh R, Melaku YA, Mensah GA, Misganaw A, Mokdad AH, Moran AE, Nawaz H, Neal B, Ngalesoni FN, Ohkubo T, Pourmalek F, Rafay A, Rai RK, Rojas-Rueda D, Sampson UK, Santos IS, Sawhney M, Schutte AE, Sepanlou SG, Shifa GT, Shiue I, Tedla BA, Thrift AG, Tonelli M, Truelsen T, Tsilimparis N, Ukwaja KN, Uthman OA, Vasankari T, Venketasubramanian N, Vlassov VV, Vos T, Westerman R, Yan LL, Yano Y, Yonemoto N, Zaki ME, Murray CJ. Global Burden of Hypertension and Systolic Blood Pressure of at Least 110 to 115 mm Hg, 1990-2015. JAMA. 2017 Jan 10;317(2):165-182. doi: 10.1001/jama.2016.19043. PMID 28097354
- [Background] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Background] Hamming I, Timens W, Bulthuis ML, Lely AT, Navis G, van Goor H. Tissue distribution of ACE2 protein, the functional receptor for SARS coronavirus. A first step in understanding SARS pathogenesis. J Pathol. 2004 Jun;203(2):631-7. doi: 10.1002/path.1570. PMID 15141377
- [Background] Ferrario CM, Jessup J, Chappell MC, Averill DB, Brosnihan KB, Tallant EA, Diz DI, Gallagher PE. Effect of angiotensin-converting enzyme inhibition and angiotensin II receptor blockers on cardiac angiotensin-converting enzyme 2. Circulation. 2005 May 24;111(20):2605-10. doi: 10.1161/CIRCULATIONAHA.104.510461. Epub 2005 May 16. PMID 15897343
- [Background] Ocaranza MP, Godoy I, Jalil JE, Varas M, Collantes P, Pinto M, Roman M, Ramirez C, Copaja M, Diaz-Araya G, Castro P, Lavandero S. Enalapril attenuates downregulation of Angiotensin-converting enzyme 2 in the late phase of ventricular dysfunction in myocardial infarcted rat. Hypertension. 2006 Oct;48(4):572-8. doi: 10.1161/01.HYP.0000237862.94083.45. Epub 2006 Aug 14. PMID 16908757
- [Background] Ishiyama Y, Gallagher PE, Averill DB, Tallant EA, Brosnihan KB, Ferrario CM. Upregulation of angiotensin-converting enzyme 2 after myocardial infarction by blockade of angiotensin II receptors. Hypertension. 2004 May;43(5):970-6. doi: 10.1161/01.HYP.0000124667.34652.1a. Epub 2004 Mar 8. PMID 15007027
- [Background] Soler MJ, Ye M, Wysocki J, William J, Lloveras J, Batlle D. Localization of ACE2 in the renal vasculature: amplification by angiotensin II type 1 receptor blockade using telmisartan. Am J Physiol Renal Physiol. 2009 Feb;296(2):F398-405. doi: 10.1152/ajprenal.90488.2008. Epub 2008 Nov 12. PMID 19004932
- [Background] Burrell LM, Risvanis J, Kubota E, Dean RG, MacDonald PS, Lu S, Tikellis C, Grant SL, Lew RA, Smith AI, Cooper ME, Johnston CI. Myocardial infarction increases ACE2 expression in rat and humans. Eur Heart J. 2005 Feb;26(4):369-75; discussion 322-4. doi: 10.1093/eurheartj/ehi114. Epub 2005 Jan 25. PMID 15671045
- [Background] Burchill LJ, Velkoska E, Dean RG, Griggs K, Patel SK, Burrell LM. Combination renin-angiotensin system blockade and angiotensin-converting enzyme 2 in experimental myocardial infarction: implications for future therapeutic directions. Clin Sci (Lond). 2012 Dec;123(11):649-58. doi: 10.1042/CS20120162. PMID 22715807
- [Background] Walters TE, Kalman JM, Patel SK, Mearns M, Velkoska E, Burrell LM. Angiotensin converting enzyme 2 activity and human atrial fibrillation: increased plasma angiotensin converting enzyme 2 activity is associated with atrial fibrillation and more advanced left atrial structural remodelling. Europace. 2017 Aug 1;19(8):1280-1287. doi: 10.1093/europace/euw246. PMID 27738071
- [Background] Ramchand J, Patel SK, Srivastava PM, Farouque O, Burrell LM. Elevated plasma angiotensin converting enzyme 2 activity is an independent predictor of major adverse cardiac events in patients with obstructive coronary artery disease. PLoS One. 2018 Jun 13;13(6):e0198144. doi: 10.1371/journal.pone.0198144. eCollection 2018. PMID 29897923
- [Background] Kuba K, Imai Y, Rao S, Gao H, Guo F, Guan B, Huan Y, Yang P, Zhang Y, Deng W, Bao L, Zhang B, Liu G, Wang Z, Chappell M, Liu Y, Zheng D, Leibbrandt A, Wada T, Slutsky AS, Liu D, Qin C, Jiang C, Penninger JM. A crucial role of angiotensin converting enzyme 2 (ACE2) in SARS coronavirus-induced lung injury. Nat Med. 2005 Aug;11(8):875-9. doi: 10.1038/nm1267. Epub 2005 Jul 10. PMID 16007097
- [Background] Henry C, Zaizafoun M, Stock E, Ghamande S, Arroliga AC, White HD. Impact of angiotensin-converting enzyme inhibitors and statins on viral pneumonia. Proc (Bayl Univ Med Cent). 2018 Oct 26;31(4):419-423. doi: 10.1080/08998280.2018.1499293. eCollection 2018 Oct. PMID 30948970
- [Background] Gu Q, Burt VL, Dillon CF, Yoon S. Trends in antihypertensive medication use and blood pressure control among United States adults with hypertension: the National Health And Nutrition Examination Survey, 2001 to 2010. Circulation. 2012 Oct 23;126(17):2105-14. doi: 10.1161/CIRCULATIONAHA.112.096156. PMID 23091084
- [Background] Buczko W, Kubik A, Kucharewicz I, Chabielska E. Antithrombotic effect of captopril and enalapril in young rats. Pol J Pharmacol. 2004 Jan-Feb;56(1):97-104. PMID 15047983
- [Background] Remkova A, Kratochvilova H. Effect of the angiotensin-converting enzyme inhibitor perindopril on haemostasis in essential hypertension. Blood Coagul Fibrinolysis. 2000 Oct;11(7):641-4. doi: 10.1097/00001721-200010000-00008. PMID 11085284
- [Background] Senchenkova EY, Russell J, Esmon CT, Granger DN. Roles of Coagulation and fibrinolysis in angiotensin II-enhanced microvascular thrombosis. Microcirculation. 2014 Jul;21(5):401-7. doi: 10.1111/micc.12120. PMID 24495184
- [Background] Wojewodzka-Zelezniakowicz M, Chabielska E, Mogielnicki A, Kramkowski K, Karp A, Opadczuk A, Domaniewski T, Malinowska-Zaprzalka M, Buczko W. Antithrombotic effect of tissue and plasma type angiotensin converting enzyme inhibitors in experimental thrombosis in rats. J Physiol Pharmacol. 2006 Jun;57(2):231-45. PMID 16845228
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Background] Bateman BT, Patorno E, Desai RJ, Seely EW, Mogun H, Dejene SZ, Fischer MA, Friedman AM, Hernandez-Diaz S, Huybrechts KF. Angiotensin-Converting Enzyme Inhibitors and the Risk of Congenital Malformations. Obstet Gynecol. 2017 Jan;129(1):174-184. doi: 10.1097/AOG.0000000000001775. PMID 27926639
- [Background] Moretti ME, Caprara D, Drehuta I, Yeung E, Cheung S, Federico L, Koren G. The Fetal Safety of Angiotensin Converting Enzyme Inhibitors and Angiotensin II Receptor Blockers. Obstet Gynecol Int. 2012;2012:658310. doi: 10.1155/2012/658310. Epub 2011 Dec 13. PMID 22203847
- [Background] Chow SC, Shao J, Wang H. Sample Size Calculations in Clinical Research. 2nd Edition ed. New York: Dekker; 2008.
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324
- [Background] PASS 16 Power Analysis and Sample Size Software. NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass. 2018.
- [Background] Willan AR, Pater JL. Carryover and the two-period crossover clinical trial. Biometrics. 1986 Sep;42(3):593-9. PMID 3567292
- [Background] Brown BW Jr. The crossover experiment for clinical trials. Biometrics. 1980 Mar;36(1):69-79. PMID 7370374
- [Background] GRIZZLE JE. THE TWO-PERIOD CHANGE-OVER DESIGN AN ITS USE IN CLINICAL TRIALS. Biometrics. 1965 Jun;21:467-80. No abstract available. PMID 14338679
- [Background] Laird NM, Ware JH. Random-effects models for longitudinal data. Biometrics. 1982 Dec;38(4):963-74. PMID 7168798
- [Background] Therneau TM, Grambsch PM. Modeling Survival Data: Extending the Cox Model. In: Statistics for Biology and Health. New York, NY: Springer; 2001.
- [Background] Little RJ. Modeling the drop-out mechanism in repeated-measures studies. Journal of the American Statistical Association. 1995;90:1112-1121.
- [Background] Xie X, Chen J, Wang X, Zhang F, Liu Y. Age- and gender-related difference of ACE2 expression in rat lung. Life Sci. 2006 Apr 4;78(19):2166-71. doi: 10.1016/j.lfs.2005.09.038. Epub 2005 Nov 21. PMID 16303146
- [Background] Wright JT Jr, Dunn JK, Cutler JA, Davis BR, Cushman WC, Ford CE, Haywood LJ, Leenen FH, Margolis KL, Papademetriou V, Probstfield JL, Whelton PK, Habib GB; ALLHAT Collaborative Research Group. Outcomes in hypertensive black and nonblack patients treated with chlorthalidone, amlodipine, and lisinopril. JAMA. 2005 Apr 6;293(13):1595-608. doi: 10.1001/jama.293.13.1595. PMID 15811979
- [Background] Gurwitz D. Angiotensin receptor blockers as tentative SARS-CoV-2 therapeutics. Drug Dev Res. 2020 Aug;81(5):537-540. doi: 10.1002/ddr.21656. Epub 2020 Mar 4. PMID 32129518
- [Background] Pflugfelder PW, Baird MG, Tonkon MJ, DiBianco R, Pitt B. Clinical consequences of angiotensin-converting enzyme inhibitor withdrawal in chronic heart failure: a double-blind, placebo-controlled study of quinapril. The Quinapril Heart Failure Trial Investigators. J Am Coll Cardiol. 1993 Nov 15;22(6):1557-63. doi: 10.1016/0735-1097(93)90578-o. PMID 8227822
- [Background] Beeftink MM, van der Sande NG, Bots ML, Doevendans PA, Blankestijn PJ, Visseren FL, Voskuil M, Spiering W. Safety of Temporary Discontinuation of Antihypertensive Medication in Patients With Difficult-to-Control Hypertension. Hypertension. 2017 May;69(5):927-932. doi: 10.1161/HYPERTENSIONAHA.116.08793. Epub 2017 Apr 3. PMID 28373591
- [Derived] Cohen JB, Hanff TC, William P, Sweitzer N, Rosado-Santander NR, Medina C, Rodriguez-Mori JE, Renna N, Chang TI, Corrales-Medina V, Andrade-Villanueva JF, Barbagelata A, Cristodulo-Cortez R, Diaz-Cucho OA, Spaak J, Alfonso CE, Valdivia-Vega R, Villavicencio-Carranza M, Ayala-Garcia RJ, Castro-Callirgos CA, Gonzalez-Hernandez LA, Bernales-Salas EF, Coacalla-Guerra JC, Salinas-Herrera CD, Nicolosi L, Basconcel M, Byrd JB, Sharkoski T, Bendezu-Huasasquiche LE, Chittams J, Edmonston DL, Vasquez CR, Chirinos JA. Continuation versus discontinuation of renin-angiotensin system inhibitors in patients admitted to hospital with COVID-19: a prospective, randomised, open-label trial. Lancet Respir Med. 2021 Mar;9(3):275-284. doi: 10.1016/S2213-2600(20)30558-0. Epub 2021 Jan 7. PMID 33422263

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Discontinuation Arm | Continuation Arm
Started | 77 | 75
Completed | 77 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Discontinuation Arm | Continuation Arm | Total
Number analyzed (Participants) | 77 | 75 | 152
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 62 (12) | 62 (12) | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 33 | 68
  Male | 42 | 42 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 40 | 82
  Not Hispanic or Latino | 35 | 35 | 70
  Unknown or Not Reported | 0 | 0 | 0
Hypertension [Count of Participants; unit: Participants]
  ACEI therapy (as opposed to ARB)* | 38 | 25 | 63
  Lowest recommended ACEI or ARB dose | 14 | 14 | 28
  Calcium channel blocker therapy | 26 | 20 | 46
  Diuretic therapy | 21 | 25 | 46
  β blocker therapy | 14 | 11 | 25
Diabetes [Count of Participants; unit: Participants]
  Insulin Therapy | 16 | 20 | 36
  No insulin therapy | 11 | 22 | 33
Dyslipidemia [Count of Participants; unit: Participants] | 32 | 34 | 66
Pre-existing cardiac disease [Count of Participants; unit: Participants] | 14 | 10 | 24
Ischemic heart disease [Count of Participants; unit: Participants] | 12 | 6 | 18
Heart Failure [Count of Participants; unit: Participants] | 3 | 3 | 6
Atrial fibrillation [Count of Participants; unit: Participants] | 0 | 3 | 3
Previous PE or DVT [Count of Participants; unit: Participants] — PE: pulmonary embolism DVT: deep vein thrombosis
  Participants | 3 | 1 | 4
Obstructive sleep apnea [Count of Participants; unit: Participants] | 10 | 7 | 17
Chronic pulmonary disease [Count of Participants; unit: Participants] | 17 | 9 | 26
Current Smoker [Count of Participants; unit: Participants] | 8 | 5 | 13
Illicit drug use [Count of Participants; unit: Participants] | 3 | 2 | 5
Dyspnoea [Count of Participants; unit: Participants] | 66 | 66 | 132
Cough [Count of Participants; unit: Participants] | 58 | 59 | 117
Multifocal infiltrates on chest x-ray or CT [Count of Participants; unit: Participants] | 43 | 48 | 91
Oxygen saturation [Mean (Standard Deviation); unit: % of oxygen in blood] — Taken with pulse oximeter, usually affixed onto right index finger. Measures the amount of oxygen in a subject's blood. A higher percentage is preferred.
  % of oxygen in blood | 92 (5) | 92 (8) | 92 (7)
Oxygen supplementation [Number; unit: number of subjects requiring extra O2] — Refers to the number of subjects requiring supplemental oxygen (given to maintain adequate levels of blood oxygenation).
  number of subjects requiring extra O2 | 60 | 63 | 61
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 133 (22) | 129 (19) | 131 (20)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 77 (12) | 75 (13) | 76 (12)
Heart rate [Mean (Standard Deviation); unit: bpm] | 92 (17) | 91 (16) | 91 (16)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33 (9) | 33 (7) | 33 (8)
eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 81 (25) | 83 (23) | 82 (24)
K Serum [Mean (Standard Deviation); unit: mmol/L] — K: potassium measured from subject's serum
  Normal levels range from 3.5-5.0 mmol/L
  mmol/L | 4 (0.5) | 4 (0.5) | 4 (0.5)
Leukocyte count [Mean (Standard Deviation); unit: 10^9 cells/L] | 8.9 (4.5) | 9.3 (4.3) | 9.1 (4.4)
Platelets [Mean (Standard Deviation); unit: 10^3 cells/microL] | 238 (130) | 239 (109) | 238 (119)
C reactive protein [Mean (Standard Deviation); unit: mg/dL] | 45 (77) | 48 (68) | 46 (72)
Days from admission to randomization [Mean (Standard Deviation); unit: days] | 1.5 (0.5) | 1.6 (0.9) | 1.5 (0.7)
Days from symptom onset to randomization [Mean (Standard Deviation); unit: days] | 6.8 (2.5) | 6.5 (2.3) | 6.65 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Hierarchical Composite Endpoint
Description: The primary endpoint of the trial will be a global rank based on patient outcomes according to four factors: (1) time to death, (2) the number of days supported by invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO), (3) the number of days supported by renal replacement therapy or pressor/inotropic therapy, and (4) a modified sequential Organ Failure Assessment (SOFA) score. The modified SOFA score will include the cardiac, respiratory, renal and coagulation domains of the SOFA score.
  How to interpret the rank?: patients are ranked from worst to best outcomes, such that patients with bad outcomes are ranked at the top and patients who have the best outcomes are ranked at the bottom.
Time Frame: Up to 28 days
Measure: Median (Inter-Quartile Range); unit: score on a scale (range 1 to 152)
Arm/Group | Discontinuation Arm | Continuation Arm
Number analyzed (Participants) | 77 | 75
score on a scale (range 1 to 152) | 81 [38 to 117] | 73 [40 to 110]

2. Secondary Outcome: All-Cause Death
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinuation Arm | Continuation Arm
Number analyzed (Participants) | 77 | 75
Participants | 10 | 11

3. Secondary Outcome: Length of Hospital Stay
Description: This outcome measurement looked at the median length of hospitalization.
Time Frame: Up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Discontinuation Arm | Continuation Arm
Number analyzed (Participants) | 77 | 75
days | 5 [3 to 10] | 6 [3 to 11]

4. Secondary Outcome: Length of ICU Stay, Invasive Mechanical Ventilation or Extracorporeal Membrane Oxygenation
Time Frame: Up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Discontinuation Arm | Continuation Arm
Number analyzed (Participants) | 77 | 75
days | 15 [6 to 27] | 13 [6 to 17]

5. Secondary Outcome: AUC SOFA
Description: The Area Under the Curve of the modified SOFA (AUC SOFA) from daily measurements, weighted to account for the shorter observation period among patients who die in-hospital.
  How to interpret the AUC SOFA?: a higher area indicates more severe disease and/or longer hospitalization.The range is 0.1 to 377.3.
Time Frame: Up to 28 days
Measure: Median (Inter-Quartile Range); unit: units on a scale (SOFA x days)
Arm/Group | Discontinuation Arm | Continuation Arm
Number analyzed (Participants) | 77 | 75
units on a scale (SOFA x days) | 7 [2 to 20] | 12 [3 to 23]

6. Other Pre Specified Outcome: Intensive Care Unit Admission or Respiratory Failure Requiring Mechanical Ventilation.
Description: Need to be transferred to an intensive care unit or to supported by a breathing machine
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinuation Arm | Continuation Arm
Number analyzed (Participants) | 77 | 75
Participants | 14 | 16

7. Other Pre Specified Outcome: Hypotension Requiring Vasopressors, Inotropes or Mechanical Hemodynamic Support
Description: Hypotension Requiring Vasopressors, inotropes or mechanical hemodynamic support (ventricular assist device or intra-aortic balloon pump).
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinuation Arm | Continuation Arm
Number analyzed (Participants) | 77 | 75
Participants | 8 | 9

ADVERSE EVENTS:
Time Frame: until hospital discharge or up to 28 days if participant were discharged prior to this time point
Description: The research team kept a log of all adverse events in the trial. A medically-qualified investigator assessed all AEs.
  The definition of adverse events and Serious Adverse Events (SAE) is presented in detail in the study protocol, available in this clinicaltrials.gov record (protocol sections 5.2 and 5.3)
Arm/Group | Discontinuation Arm | Continuation Arm
All-Cause Mortality (participants affected / at risk) | 10/77 | 11/75
Serious Adverse Events (participants affected / at risk) | 28/77 | 29/75
Other Adverse Events (participants affected / at risk) | 0/77 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Discontinuation Arm (N=77) | Continuation Arm (N=75)
Delirium or encephalopathy (Investigations) | 8 | 2
New or worsening congestive heart failure (Cardiac disorders) | 1 | 2
Myocarditis (Cardiac disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Pulmonary embolism or deep vein thrombosis (Vascular disorders) | 1 | 4
Acute arrhythmia (Cardiac disorders) | 3 | 6
Acute kidney injury, defined as >2-fold increase in creatinine (Renal and urinary disorders) | 3 | 3
Acute kidney injury requiring renal replacement therapy (Renal and urinary disorders) | 1 | 2
Hypotension requiring hemodynamic support (Vascular disorders) | 8 | 9
Invasive mechanical ventilation (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Worsening dyspnoea or acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 13 | 17
ICU transfer (General disorders) | 14 | 16
All-cause death (General disorders) | 10 | 11

LIMITATIONS AND CAVEATS:
Limitations of the study include (1) small sample size; (2) we did not control participant ACEI or ARB dosing or other medication exposures during the trial; (3) Although outcome adjudicators were masked to the randomly assigned groups when determining clinical endpoints, providers caring for the patients were aware of the group the patient was assigned to. It is possible that the open-label nature of the study might have introduced information bias or influenced provider behavior.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT04338009/Prot_SAP_000.pdf